CLINICAL TRIAL: NCT03998306
Title: Influence of the Probiotic Streptococcus Salivarius K12 on Dental Health in Children With Early Childhood Caries
Brief Title: Probiotics in Children With Early Childhood Caries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KB/202/2017
Record Dates: First submitted 2019-04-15; First posted 2019-06-26 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-04

CONDITIONS: Dietary Supplement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): A half of the participants will be randomly allocated to the probiotics group. They will receive probiotic lozenge before falling asleep for12 weeks. They will receive hygienic and dietetic instructions. examination will be conducted before study and after 12 weeks.
  Interventions: Dietary Supplement: Experimental: Probiotics
- CONTROL (Sham Comparator): no intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Dietary Supplement: Experimental: Probiotics — the participants will receive probiotic lozenge before falling asleep for 12 weeks.
  the participants will receive dietetic and hygienic instructions
  Arms: Probiotics
Other: No intervention — No intervention
  Arms: CONTROL

SUMMARY:
The purpose of this study is to determine if probiotic lozenges taken once a day before bedtime for twelve weeks can decrease the numbers of Streptococcus mutans

DETAILED DESCRIPTION:
Streptococcus salivarius is one of the commensal bacteria of the mouth and the main component of biofilm. Research indicates that some microorganisms present in plaque, which until recently were considered not to cause caries, including Streptococcus salivarius, present in the supragingival microbiome, can also cause tooth decay.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy children aged 3-6;
* recognized caries of early childhood, dmf> 1,
* lack of active caries and inflammation of the mouth
* CFU> 105 / ml Streptococcus mutans
* a minimum of one-month period from: the last antibiotic therapy, probiotic use, professional fluoride prophylaxis or supervised tooth brushing with fluoride preparations, the use of fluoride toothpaste, not using xylitol, written consent of parents / legal guardians for participation in research.

Exclusion Criteria:

chronic diseases and chronically taken medicines in the past,

* planned change of residence during the year,
* age below 3 and above 6 years,
* healthy teeth, dmf = 0,
* CFU <105 / ml Streptococcus mutans
* Patient during antibiotic therapy, probiotic use, professional fluoride prophylaxis or supervised tooth brushing with fluoride preparations
* no toothpaste with fluoride
* using xylitol
* lack of written consent of parents / legal guardians for participation in research.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Changing the amount of carcinogenic bacteria Streptococcus mutans in intervention group based on bacterial test counting number of Colony Forming Units | 12 weeks
  During control test saliva will be applied to the medium for identification and detailed quantification of Streptococcus mutans bacteria. After the incubation, the number of bacteria will be expressed - taking into account the degree of saliva dilution - as the number of colony-forming unit (CFU) in 1 ml of saliva. colony forming unit CFU in intervention and control groups. Bacterial tests will be used to assess this outcome measure. We expect decrement of amount of cariogenic bacteria in intervention group

CONTACTS AND LOCATIONS:
Locations (1):
- Dorota Olczak-Kowalczyk, Warsaw, Warsaw, 18 Miodowa Saint, Poland